CLINICAL TRIAL: NCT02277301
Title: Mellow Babies - a Pilot Waiting List Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: South Eastern Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Dr Lucy Thompson, Senior Research Fellow, University of Aberdeen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2/033/14
Record Dates: First submitted 2014-10-24; First posted 2014-10-29 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Mothers Who Have Been Referred for Parenting Support
Keywords: Pilot study; Randomised Controlled Trial; Parenting; Paediatrics; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mellow Babies (Experimental): Mellow Babies is a group day programme, run one day a week over 14 weeks with a joint focus on maternal wellbeing and the parentinfant interaction: transport and crèche facilities are provided.The focus is to: (a) explicitly enhance close mother-infant attunement, using a combination of baby-massage, interaction coaching and infant focussed speech; and (b) offer mothers support for their own distress. Mellow Babies is an intervention designed for mothers with substantial problems in their relationships with their infants. Typically, participating mothers have mental health difficulties, problem drug use, learning difficulties, forensic issues or they may have children already looked after by the local authority.
  Interventions: Behavioral: Mellow Babies
- Care as Usual (No Intervention): Routine care received by mothers with substantial problems in their relationships with their infants. Typically, participating mothers have mental health difficulties, problem drug use, learning difficulties, forensic issues or they may have children already looked after by the local authority.

INTERVENTIONS:
Behavioral: Mellow Babies — Mellow Babies is an intervention designed for mothers with substantial problems in their relationships with their infants. Typically, participating mothers have mental health difficulties, problem drug use, learning difficulties, forensic issues or they may have children already looked after by the local authority.
  Other Names: Mellow Parenting
  Arms: Mellow Babies

SUMMARY:
This is a mixed-methods study centred on a prospective randomised openlabel blinded endpoint (PROBE) pilot clinical trial with a waitinglist control group. The study will be conducted in three areas of Northern Ireland: Lisburn, North Down & Ards, and Downpatrick. At least 50 women with infants under 13 months old will be recruited during August/September 2014.

DETAILED DESCRIPTION:
Psychologically informed very early intervention programmes across the ante- and postnatal period have shown promise in delivering cost-effective long term positive outcomes. There is robust support for the view that early intervention to prevent and manage difficulties in the parent-infant relationship may produce long-term benefits such as reduction in rates of criminality, substance abuse and educational underachievement. A meta-analysis of sensitivity and attachment interventions in early childhood has shown that the most effective interventions use a moderate number of sessions (n=5-16) and are focussed on parental sensitivity.

Although Mellow Parenting interventions (Mellow Babies is probably the best-evidenced) are quite widely used in a number of countries, no definitive randomised trials have been carried out. To date there has been a single small waiting list trial suggesting improvement in maternal mood and mother-child interaction, We aim to inform the design of a definitive RCT with a waiting-list control trial with adequate power to estimate an effect size.

This is a parallel randomised open-label blinded end-point (PROBE) clinical trial with a waiting-list control group. The study will be conducted in three areas: Lisburn, North Down & Ards, and Downpatrick. At least 50 women with infants under 18 months old will be recruited in September 2014. Participating women will be given information on the study, in particular being informed that participation would involve either receiving the intervention the following month or after a delay of 20 weeks. Signed consent (which will include consent to follow up after one year, beyond the timespan of this study) will be sought after an interval of at least 24 hours to allow the women to arrive at an informed decision.

ELIGIBILITY:
Inclusion Criteria:

Mothers of infants aged less then 13 months who have been referred for parenting support by the health or social care services.

Exclusion Criteria:

Those unable to complete research assessments (due to literacy or language issues).

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Mellow Parenting Observation System (MPOS). | 16-18 weeks
  MPOS, is an event sampled observational system in which the rate of positive and negative parenting behaviours is calculated.

SECONDARY OUTCOMES:
The Adult Wellbeing Scale (Snaith et al 1978) | 16-18 weeks
  The Adult Wellbeing Scale is based on the Hospital Anxiety and Depression Scale which is used to determine the levels of anxiety and depression that a patient is experiencing.

OTHER OUTCOMES:
The Edinburgh Postnatal Depression Scale (Cox et al 1987) - | 16-18 weeks
  The Edinburgh Postnatal Depression Scale is the standard clinical screening tool for postnatal depression, widely used by health visitors.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Thompson, BA PhD MPH, Principal Investigator — University of Aberdeen
Locations (1):
- Lisburn Health Centre, Lisburn, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thompson L, Wilson P. Mellow Babies: A Randomised Feasibility Trial of an Intervention to Improve the Quality of Parent-Infant Interactions and Parental Mental Wellbeing. Children (Basel). 2024 Apr 24;11(5):510. doi: 10.3390/children11050510. PMID 38790505